CLINICAL TRIAL: NCT05437679
Title: ANG-015 / MLU-3 (CHARTER Study): Characterization of Circulating Tumor Cells Isolated Using the Parsortix® System in High Risk and Early Metastatic Prostate Cancer Patients
Brief Title: Characterization of Circulating Tumor Cells (CTCs) in High Risk and Early Metastatic Prostate Cancer Patients Using Parsortix® System
Acronym: CHARTER
Status: Terminated | Type: Observational
Why Stopped: Futility (slow enrollment)
Sponsor: Angle plc (Industry)
Collaborators: MidLantic Urology, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANG-015 / MLU-3
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: High Risk Prostate Carcinoma; Biochemically Recurrent Prostate Carcinoma; Castration-resistant Prostate Cancer; Prostate Cancer
Keywords: surveillance; circulating tumor cells; PETCT; PSMA; Axumin; Parsortix; next generation imaging
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected, and the following will be isolated from the whole blood samples: serum, plasma, cells (e.g., CTCs, white blood cells, etc.), circulating cell free DNA, DNA and RNA from isolated cells, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Active Surveillance (AS) Controls: Patients with low or very low risk prostate cancer who have been on active surveillance for 5 or more years with a stable PSA or on active surveillance for 2 or more years with negative multiparametric MRI (mpMRI) or mpMRI with a fusion biopsy(ies) confirming low risk disease.
  Interventions: Other: Blood collection
- High Risk Localized Prostate Cancer (HRLPC): Men with high-risk localized prostate cancer, defined as stage pT3a or Gleason score greater than or equal to 8 and/or pre-prostatectomy PSA of greater than or equal to 20 ng/mL.
  Interventions: Other: Blood collection
- Biochemically Recurrent Localized Prostate Cancer (BCRLPC): Systemic and/or hormonal treatment naive men with localized prostate cancer (pathological stages pT2, pT3a or pT4 with TNM N0 or N1 and M0 disease) who have clinical suspicion of biochemical recurrence 2 - 5 months following radical prostatectomy and are scheduled to undergo NGI (i.e., Axumin® or PSMA PETCT) within the next 45 days or have already undergone NGI within the past 45 days.
  Interventions: Other: Blood collection
- Non-Metastatic Castration-Resistant Prostate Cancer (NMCRPC): Patients with evidence of non-metastatic castration-resistant prostate cancer (i.e. localized prostate cancer patients with clinical symptoms of disease progression and/or evidence of a rising PSA following hormone therapy) who are scheduled to undergo NGI (i.e., Axumin® or PSMA PETCT) within the next 45 days or have already undergone NGI within the past 45 days and who have not started a new therapy for treatment of their castration-resistant prostate cancer.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Peripheral blood will be collected from each subject at a single time point and data will be collected from a review of each subject's medical records.
  Other Names: Data collection

SUMMARY:
This study is designed to evaluate the presence and numbers of circulating tumor cells (CTCs) and cancer related gene expression levels in subjects with localized high-risk prostate cancer (HRLPC) and from subjects with non-metastatic disease experiencing biochemical recurrence and castration-resistance (BCRLPC and NMCRPC groups, respectively) who are about to undergo next generation imaging (NGI, such as Axumin® or PSMA PETCT). The investigators will also evaluate subjects with localized indolent prostate cancer who are on active surveillance (AS) as a control population. The CTC and gene expression results will be evaluated for association with disease state and progression and survival.

DETAILED DESCRIPTION:
Patients who meet the eligibility criteria and provide written informed consent will be enrolled into the study. The four (4) groups of patients to be enrolled into the study will consist of: 1) men with low risk localized prostate cancer (LPC) on active surveillance (AS control group), 2) treatment naïve men with high risk LPC (HRLPC) who are 2 - 5 months out after having a radical prostatectomy, 3) treatment naïve men with biochemically recurrent LPC (BCRLPC) who are about to or have recently undergone next generation imaging [NGI] (i.e. Axumin® or PSMA PETCT), and men with non-metastatic castration resistant prostate cancer (NMCRPC) who are about to or have recently undergone NGI (i.e. Axumin® or PSMA PETCT). The goal is to enroll a total of 25 evaluable patients into each study group (HRLPC, BCRLPC, NMCRPC and AS) and collect up to ~29mL of blood from each patient as a single timepoint for evaluation. HRLPC patients will have blood draw 2 - 5 months following their radical prostatectomy procedure, BCRLPC and NMCRPC patients will have their blood drawn within 45 days prior to or after their scheduled NGI study and prior to initiation of a new treatment for their disease, and AS patients will have their blood drawn either after having a stable PSA for greater than 5 years or greater than 2 years after having a biopsy confirming low risk disease. All patients will be followed for up to 2 years after enrollment for disease progression and survival status.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 18 years of age;
* ECOG status of 0 - 2;
* Signed informed consent;
* HRLPC cohort (n=25):

  * Clinical diagnosis of HRLPC, defined as stage pT3a or Gleason score >8 and/or pre-prostatectomy PSA >20 ng/mL;
  * 2-5 months post-radical prostatectomy;
  * Treatment naïve (i.e. have not received any systemic and/or hormonal therapy since the time of their radical prostatectomy).
* BCRLPC cohort (n=25):

  * Patients with localized prostate cancer (pathological stages pT2, pT3a, pT3b or pT4 with TNM N0 or N1 and M0 disease) who have clinical suspicion of biochemical recurrence following a radical prostatectomy;
  * Have been pre-authorized by insurance to undergo next generation imaging (NGI, such as Axumin® or PSMA PETCT) within the next 45 days or have already undergone NGI within the past 45 days;
  * Treatment naïve (i.e. have not received any systemic and/or hormonal therapy since the time of their radical prostatectomy).
* NMCRPC cohort (n=25):

  * Patients with evidence of non-metastatic castration-resistant prostate cancer (i.e. localized prostate cancer patients with clinical symptoms of disease progression and/or evidence of a rising PSA following hormone therapy);
  * Have been pre-authorized by insurance to undergo NGI (i.e. Axumin® or PSMA PETCT) within the next 45 days or have already undergone NGI within the past 45 days;
  * Have not started a new therapy for the treatment of their castration-resistant prostate cancer.
* Control cohort (n=25):

  * Patients with low or very low risk prostate cancer who have been on active surveillance (AS) for 5 or more years with a stable PSA or on active surveillance for 2 or more years with negative multiparametric magnetic resonance imaging (mpMRI) or mpMRI with a fusion biopsy confirming low risk disease.

Exclusion Criteria:

* Documented evidence of brain metastases;
* ECOG status of 3 or greater;
* Unable to provide informed consent or a high risk that the patient may not comply with the protocol requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated within MidLantic Urology's (MLU's) clinical network (located in southeast Pennsylvania), will be evaluated for eligibility and invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
CTC number and phenotype | Baseline
  The population of cells captured from the peripheral blood samples by the Parsortix system will be evaluated using cytological and/or immunofluorescent staining methods to determine the numbers and phenotypes of any rare cells present (e.g., epithelial and/or mesenchymal CTCs, megakaryocytes, etc. alone and/or in clusters). The numbers and phenotypes of any rare cells present will be evaluated for association with the patient disease state (e.g., study group), the presence of metastatic disease as determined by NGI, and disease progression and/or survival (for up to two years following enrollment).
CTC genotype | Baseline
  DNA and/or RNA will be isolated from the population of cells captured from the peripheral blood samples by the Parsortix system and will be evaluated using molecular methods (e.g. multiplex gene expression, mutational analysis, sequencing, etc.) to determine the genotype(s) of the harvested cells. The genotype(s) of any rare cells present will be evaluated for association with the patient disease state (e.g., study group), the presence of metastatic disease as determined by NGI, and disease progression and/or survival (for up to two years following enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Moreno, MD, Principal Investigator — MidLantic Urology, LLC
Locations (2):
- United States (2):
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - MidLantic Urology, Pottstown, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be shared with other researchers.

REFERENCES:
- [Background] Moreno JG, Gomella LG. Evolution of the Liquid Biopsy in Metastatic Prostate Cancer. Urology. 2019 Oct;132:1-9. doi: 10.1016/j.urology.2019.06.006. Epub 2019 Jun 14. PMID 31207303
- [Background] Miller MC, Robinson PS, Wagner C, O'Shannessy DJ. The Parsortix Cell Separation System-A versatile liquid biopsy platform. Cytometry A. 2018 Dec;93(12):1234-1239. doi: 10.1002/cyto.a.23571. Epub 2018 Aug 14. PMID 30107082
- See also: MidLantic Urology, LLC — https://midlanticurology.com/
- See also: ANGLE plc — https://angleplc.com/